CLINICAL TRIAL: NCT04249804
Title: Intravenous Infusion Versus Intrathecal Injection of Magnesium Sulfate for Prevention of Postspinal Shivering During Lower Limb Fracture Surgery. A Randomized Comparative Study
Brief Title: the Use of Magnesium Sulfate for Prevention of Postspinal Shivering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-261-2019
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Prevention of Postspinal Shivering
Keywords: Magnesium Sulfate - postspinal shivering -intrathecal - infusion
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated to Groups ([T], Intrathecal MgSo4 and [M], IV infusion MgSo4 groups) on the basis of computer-generated random numbers. Patients belonging to Group T (n = 45) will receive 50 mg intrathecal MgSo4 added to 0.5% hyperbaric bupivacaine [131],while those belonging to Group M (group, n = 45) will receive IV magnesium sulfate 50 mg/kg in 100 mL isotonic saline over 20 min as a bolus then 2 mg/kg/h infusion using a separate infusion set after administering spinal anesthesia.
  Axillary temperature and grades of shivering will be noted every 10 min by the same anesthesiologist who performed the spinal anesthesia using Crossley and Mahajan scale,[8] If grade III, IV shivering persisted for >10 min pethidine 25 mg IV will be administered as a rescue drug and number of patients required rescue drug will be recorded.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrathecal Mg group (Experimental): 45 patients will receive 50 mg intrathecal MgSo4 added to 0.5% hyperbaric bupivacaine
  Interventions: Drug: Magnesium Sulfate 1000 MG
- IV Mg infusion group (Experimental): 45 patients will receive IV magnesium sulfate 50 mg/kg in 100 mL isotonic saline over 20 min as a bolus then 2 mg/kg/h infusion using a separate infusion set after administering spinal anesthesia
  Interventions: Drug: Magnesium Sulfate 1000 MG
- control (No Intervention): 0.5% heavy bupivacaine in the spinal with no additives

INTERVENTIONS:
Drug: Magnesium Sulfate 1000 MG — intrathecal versus IV infusion of Magnesium sulfate for prevention of postspinal shivering
  Arms: IV Mg infusion group; Intrathecal Mg group

SUMMARY:
Shivering is an unpleasant experience after spinal anesthesia. Shivering is defined as an involuntary, repetitive activity of skeletal muscles. The mechanisms of shivering in patients undergoing surgery are mainly intraoperative heat loss, increased sympathetic tone, pain, and systemic release of pyrogens. Spinal anesthesia significantly impairs the thermoregulation system by inhibiting tonic vasoconstriction, which plays a significant role in temperature regulation. Spinal anesthesia also causes redistribution of core heat from the trunk (below the block level) to the peripheral tissues. These two effects predispose patients to hypothermia and shivering. The median incidence of shivering related to regional anesthesia observed in a review of 21 studies is 64.4%. Shivering increases oxygen consumption, lactic acidosis, carbon dioxide production, and metabolic rate by up to 400%. Therefore, shivering may cause problems in patients with low cardiac and pulmonary reserves. The best way to avoid these intraoperative and postoperative shivering-induced increases in hemodynamic and metabolic demands is to prevent shivering in the first place. Although magnesium is among several pharmacological agents used for the treatment of shivering, its effects on prevention of shivering during central neuraxial blockade have not been evaluated to date. Henceforth, the aim of this study was to evaluate the effect of magnesiume on shivering during spinal anesthesia.

Aim:

to compare the efficacy of intravenous versus intrathecal magnesium sulphate for prevention of post spinal shivering in adult patients undergoing elective lower limb orthopedic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-45 years old
* Both genders
* ASA I, II

Exclusion Criteria:

* Patients with hemodynamic instability
* cardiopulmonary
* renal , liver disease
* hypo or hyperthyroidism
* cerebrovascular insufficiency
* coagulation defects
* those with psychiatric disorder
* patients receiving vasoactive drugs or beta blockers
* BMI > 35
* allergic to study drug
* height <160 cm or >190 cm
* basal body temperature >38°C or <36°C
* those who received blood transfusion or >2000 mL fluid intra-operatively
* surgery duration > 3 hours

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
incidence of postspinal shivering | up to 5 months
  the efficacy of the use of MgSo4 IV infusion versus intrathecal injection in decreasing the incidence of postspinal shivering using Crossley and Mahajan scale which is 0, no shivering; 1, piloerection or peripheral vasoconstriction (cyanosis) but no visible shivering; 2, muscular activity in only one muscle group; 3, muscular activity in more than one muscle group but not generalized shivering; and 4, shivering involving the whole body

CONTACTS AND LOCATIONS:
Locations (1):
- anesthesia department at Cairo University, Cairo, Elmanial, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: January to May 2020

REFERENCES:
- [Background] 1. Frank S.M., Higgins M.S., Breslow M.J., et al. The catecholamine, cortisol, and hemodynamic responses to mild perioperative hypothermia: a randomized clinical trial Anesthesiology,1995, 82:83-93. 2. Crowley LJ, Buggy DJ .Shivering and neuraxial anesthesia.Reg Anesth Pain Med. 2008 May-Jun;33(3):241-52. doi: 10.1016/j.rapm.2007.11.006. 3. Mizobe T., Nakajima Y., Sunaguchi M., et al.Clonidine produces a dose-dependant impairment of baroreflex-mediated thermoregulatory responses to positive end-expiratory pressure in anesthetized humans.BJA, 2005, 94:536-541 4. Witte J. De, Sessler D.I.Perioperative shivering: physiology and pharmacology.Anesthesiology, 2002,96:467-484 5. Eberhart LH, Döderlein F, Eisenhardt G, et al Independent risk factors for postoperative shivering. Anesth Analg,2005, 101:1849-1857. 6. Lyons B, Power C, Casey W.Postanaesthesia shivering in children. Anaesthesia 1996.51: 442-445. 7. Hull D, Smales . Heat production in the newborn. In: Sinclair JC (eds.) Temperature Regulation and Energy Metabolism in the Newborn. Grune& Stratton, New York.1978 46:129-156 8. Crossley AW, Mahajan RP. The intensity of postoperative shivering is unrelated to axillary temperature. Anaesthesia 1994,49:205-207 9. P. Kranke, L.H. Eberhart, N. Roewer, M.R. TramerSingle-dose parenteral pharmacological interventions for the prevention of postoperative shivering: a quantitative systematic review of randomized controlled trials Anesth Analg, 2004, 99 :718-727 10. T. Ikeda, T. Kazama, D.I. Sessler, et al.Induction of anesthesia with ketamine reduces the magnitude of redistribution hypothermia.Anesth Analg, 2001,93: 934-938 11. S. Kizilirmak, S.E. Karakas, O. Akca, et al.Magnesium sulfate stops postanesthetic shivering.Ann NY Acad Sci, 1997813: 799-806 12. R.M. Zweifler, M.E. Voorhees, M.A. Mahmood, M. Parnell.Magnesium sulfate increases the rate of hypothermia via surface cooling and improves comfort.Stroke, 2004,35:2331-2334 13. D.B. Cotton, M. Hallak, C. Janusz, S.M. Irtenkauf, R.F. BermanCentral anticonvulsant effects of magnesium sulfate on N-methyl-D-aspartate-induced seizures.Am J Obstet Gynecol, 1993,168:974-978 14. C. Lee, X. Zhang, W.F. Kwan.Electromyographic and mechanomyographic characteristics of neuromuscular block by magnesium sulphate in the pig.Br J Anaesth, 1996,76:278-283 15. V. Rukshin, P.K. Shah, B. Cercek, A. Finkelstein, V. Tsang, S. Kaul.Comparative antithrombotic effects of magnesium sulfate and the platelet glycoprotein IIb/IIIa inhibitors tirofiban and eptifibatide in a canine model of stent thrombosis.Circulation, 2002,105:1970-1975 16. Gozdemir M, Usta B, Demircioglu RI, Muslu B, Sert H, Karatas OF. Magnesium sulfate infusion prevents shivering during transurethral prostatectomy with spinal anesthesia: a randomized, double-blinded, controlled study. J Clin Anesth. 2010,22:184-189.